CLINICAL TRIAL: NCT06853925
Title: A Pilot Randomized Controlled Trial of the Use of a Website About Radioactive Iodine Symptom Management in Patients With Thyroid Cancer
Brief Title: Testing a Web-based Intervention for Radioactive Iodine Symptom Management to Improve Health-related Quality of Life Among Differentiated Thyroid Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Alaina Carr, Assistant Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 00008478
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Neoplasms
Keywords: symptom burden; self efficacy; feasibility studies; internet-based intervention; pilot projects; neoplasms; radioactive iodine treatment; iodine radioisotopes; health-related quality of life; informational needs
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (Other): The American Cancer Society (ACS) website on Radioactive Iodine (Radioiodine)Therapy for Thyroid Cancer is the TAU comparison. This website is a reputable and trusted source of information about cancer, with relevant content and web availability. Using the ACS website allows participants in both groups to receive information (addressing ethical concerns) through a website (similar delivery mode for information).
  Interventions: Other: Treatment as Usual (TAU)
- Radioactive Iodine Support (RAI Support) (Experimental): RAI Support consists of multimedia content (images, videos, text, audio, and infographics across different website pages) that is written at an 8th grade reading level. RAI Support uses patient materials that are visually diverse to appeal to patients from different racial and ethnic backgrounds and inclusion of all genders. RAI Support users can access short (~3 minutes or less) clinician-approved symptom management education videos and follow clinician-led video-guided activities such as nutrition management for dry mouth. In addition, RAI Support contains infographic pages about specific symptoms of RAI (e.g., salivary, lacrimal, and nasal symptoms with strategies for symptom management) and a resources page consisting of a printable treatment summary and survivorship plan to bring to provider appointments and access to evidence-based stress-management resources such as relaxation recordings.
  Interventions: Behavioral: Radioactive Iodine Support (RAI Support)

INTERVENTIONS:
Behavioral: Radioactive Iodine Support (RAI Support) — RAI Support consists of multimedia content (images, videos, text, audio, and infographics across different website pages) that is written at an 8th grade reading level. RAI Support uses patient materials that are visually diverse to appeal to patients from different racial and ethnic backgrounds and inclusion of all genders. RAI Support users can access short (~3 minutes or less) clinician-approved symptom management education videos and follow clinician-led video-guided activities such as nutrition management for dry mouth. In addition, RAI Support contains infographic pages about specific symptoms of RAI (e.g., salivary, lacrimal, and nasal symptoms with strategies for symptom management) and a resources page consisting of a printable treatment summary and survivorship plan to bring to provider appointments and access to evidence-based stress-management resources such as relaxation recordings.
  Arms: Radioactive Iodine Support (RAI Support)
Other: Treatment as Usual (TAU) — The American Cancer Society (ACS) website on Radioactive Iodine (Radioiodine)Therapy for Thyroid Cancer is the TAU comparison. This website is a reputable and trusted source of information about cancer, with relevant content and web availability. Using the ACS website allows participants in both groups to receive information (addressing ethical concerns) through a website (similar delivery mode for information).
  Arms: Treatment as usual (TAU)

SUMMARY:
The goal of this clinical trial is to learn if adult patients diagnosed with differentiated thyroid cancer can easily use and benefit from an online tool aimed to provide patients with educational resources and symptom management strategies to improve their quality of life after radioactive iodine (RAI) treatment. The main questions it aims to answer are:

1. Can patients easily use and benefit from the RAI Support intervention?
2. Does RAI Support improve health-related quality of life (overall well-being) compared to usual care?

This research will help test better digital tools to support thyroid cancer survivors in managing their health after RAI treatment.

Researchers will compare RAI Support to treatment as usual (a publicly available informational website about thyroid cancer) to see if RAI Support works to improve patients' overall well-being.

Participants will:

1. Receive access to RAI Support or an informational website (treatment as usual) for four weeks.
2. Use the assigned website once a week for up to four weeks.
3. Complete two online questionnaires (an initial questionnaire and a final questionnaire after four weeks of using the assigned website) about symptoms related to RAI treatment, mood, and confidence in managing symptoms.
4. Complete an optional 60 minute virtual interview about your experiencing using the assigned website.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older (papillary or follicular carcinoma)
* Diagnosed with differentiated thyroid cancer
* Received radioactive iodine (RAI) treatment less than or equal to three years ago.
* Mild to moderate symptoms of RAI
* Able to provide informed consent in English
* Access to a computer, tablet, or smartphone with internet connectivity

Exclusion Criteria:

* A condition that precludes providing informed consent or completing study procedures (cognitive or psychiatric condition, hearing problems) as identified by the patient's physician or as assessed by a trained study team member.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Retention and Engagement) | 4 weeks
  Feasibility is defined by at least 86% of patients are retained and complete the 4-week post-assessment. Feasibility is also defined as greater or equal to 70% RAI Support engagement rate (greater or equal to 3/4 website sections).
Acceptability (Quantitative) | 4 weeks
  Acceptability will be assessed using the Acceptability of Intervention Measure (AIM). AIM is a 4-item questionnaire that assesses the acceptability of an intervention. Each item is on a 5-point Likert scale (1=Completely disagree; 5= Completely agree). Higher scores indicate greater acceptability.
Acceptability (Qualitative) | 4 weeks
  Acceptability will also be assessed from qualitative feedback gathered from participants in the RAI Support intervention condition. Up to 20 RAI Support completers will be asked to complete an individual exit interview with the PI or a trained study team member to elicit feedback on the helpfulness of the intervention, participant burden, barriers to intervention participation, satisfaction with components of the intervention, and satisfaction with the delivery, modality, and length of the intervention.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy- General-7 (FACT-G7; Health-related quality of life) | 4 weeks
  The Functional Assessment of Cancer Therapy- General-7 (FACT-G7) questionnaire consists of 7 items assessing the physical, emotional, and functional well-being of adult cancer patients. Each item is on a five-point Likert scale (0= Not at all; 4= Very much). Scores range from 0-28. Higher scores are indicative of better HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Alaina Carr, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Carr AL, Jenkins AM, Jonklaas J, Gabriel K, Miller K, Graves K. Patient and Provider Perspectives of a Web-based Intervention to Support Symptom Management after Radioactive Iodine Treatment for Differentiated Thyroid Cancer: Qualitative Study. JMIR Form Res. 2025 Feb 12. doi: 10.2196/60588. Online ahead of print. PMID 39937181

DOCUMENTS (1):
  • Informed Consent Form (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT06853925/ICF_002.pdf